CLINICAL TRIAL: NCT01952600
Title: Empowering Patients On Choices for Renal Replacement Therapy (Aim 1)
Acronym: EPOCH-RRT
Status: Completed | Type: Observational
Sponsor: Arbor Research Collaborative for Health (Other)
Collaborators: University of Michigan (Other); Henry Ford Health System (Other); National Kidney Foundation, United States (Other); American Association of Kidney Patients (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 110920130510
Record Dates: First submitted 2013-06-28; First posted 2013-09-30 (Estimated); Results first posted 2016-08-08 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Hemodialysis; Peritoneal Dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Chronic Kidney Disease (CKD): Patients who have advanced chronic kidney disease, but are not currently on either hemodialysis (HD) or peritoneal dialysis (PD).
- Hemodialysis (HD): Patients who have chronic kidney disease (CKD) and are currently on hemodialysis.
- Peritoneal Dialysis (PD): Patients who have chronic kidney disease (CKD) and are currently on peritoneal dialysis.

SUMMARY:
The EPOCH-RRT study seeks to fill knowledge gaps by gaining more understanding of chronic kidney disease (CKD) patients' priorities; assessing the comparative benefits of hemodialysis (HD) versus peritoneal dialysis (PD), with respect to these priorities; and providing tailored information to assist patients with identifying the best dialysis modality fit for their own unique circumstances and perspectives.

The outcomes most relevant to patients ("patient-centered") extend beyond those traditionally assessed in clinical research, with the relative importance varying across patient groups. A tailored decision aid based on these findings can improve patient decision-making processes regarding choice of dialysis modality.

DETAILED DESCRIPTION:
Empowering Patients On Choices for Renal Replacement Therapy (EPOCH-RRT)study seeks to identify factors that matter the most to patients with kidney disease and study how they are impacted by different types of dialysis. The inclusion of patients, caregivers, and patient advocacy organizations as research partners will assure that the study addresses questions of greatest relevance to patients facing the need for dialysis.

Aim One of EPOCH-RRT identifies outcomes that are most important to different groups of advanced CKD and dialysis patients through qualitative methods applied for conducting in-depth interviews.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years of age or older.
* Individuals with advanced chronic kidney disease or on dialysis (in-center, hemodialysis, or peritoneal dialysis) for at least three months.

Exclusion Criteria:

* Individuals under 18 years of age.
* Individuals unable to provide informed consent.
* Individuals who do not have chronic kidney disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients residing in the United States with advanced chronic kidney disease or on dialysis.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Tentori, MD, MS, Principal Investigator — Arbor Research Collaborative for Health
Locations (1):
- Arbor Research Collaborative for Health, Ann Arbor, Michigan, United States

REFERENCES:
- See also: Arbor Research Collaborative for Health is committed to improving patient care through research that shapes medical policies and practice. — http://www.arborresearch.org/
- See also: The University of Michigan Division of Nephrology is internationally recognized for its excellence in clinical care, rich educational offerings, and diverse research programs. — http://www.med.umich.edu/intmed/nephrology/
- See also: University of Michigan Center for Managing Chronic Disease aims to build the capacity for effective chronic disease prevention and management. — http://cmcd.sph.umich.edu/
- See also: The National Kidney Foundation is a voluntary nonprofit health organization dedicated to preventing kidney disease. — http://www.kidney.org/
- See also: The American Association of Kidney Patients is dedicated to improving the lives of kidney patients and their families by helping them deal with the physical, emotional, and social impact of kidney disease. — http://www.aakp.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chronic Kidney Disease (CKD) | Hemodialysis (HD) | Peritoneal Dialysis (PD)
Started | 80 | 90 | 45
Completed | 65 | 77 | 38
Not Completed | 15 | 13 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Kidney Disease (CKD) | Hemodialysis (HD) | Peritoneal Dialysis (PD) | Total
Number analyzed (Participants) | 65 | 77 | 38 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 55 | 31 | 117
  >=65 years | 34 | 22 | 7 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.40 (56.14) | 56.14 (16.65) | 50.37 (14.81) | 57.54 (16.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 36 | 20 | 99
  Male | 22 | 41 | 18 | 81
Region of Enrollment [Number; unit: participants]
  United States | 65 | 77 | 38 | 180

OUTCOME MEASURES:

1. Primary Outcome: Factors That Are Most Important to Patients
Description: Differences in factors most important to patients were compared across chronic kidney disease, hemodialysis, and peritoneal dialysis patients.
Time Frame: Baseline
Measure: Number; unit: % of patients
Arm/Group | Chronic Kidney Disease (CKD) | Hemodialysis (HD) | Peritoneal Dialysis (PD)
Number analyzed (Participants) | 65 | 77 | 38
% of patients
  Keeping as much independence as possible | 98 | 93 | 97
  Quality and quantity of life | 100 | 89 | 92
  Flexibility in daily schedule | 90 | 0 | 94
  Important to do dialysis at home | 67 | 0 | 89
  Planned schedule at dialysis center | 68 | 76 | 0
  Safer to do dialysis at a medical place | 55 | 74 | 0
  Ability to go to school and work | 43 | 0 | 71
  Concern about the way you look | 43 | 32 | 42
  Spending time with patients at dialysis center | 21 | 52 | 0
  Worry about how dialysis will affect others | 43 | 33 | 29

ADVERSE EVENTS:
Arm/Group | Chronic Kidney Disease (CKD) | Hemodialysis (HD) | Peritoneal Dialysis (PD)
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/77 | 0/38
Other Adverse Events (participants affected / at risk) | 0/65 | 0/77 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No